CLINICAL TRIAL: NCT04526652
Title: Evaluating Stress Response and Anxiety Score in Paediatric Patients Sedated With Intranasal Dexmedetomidine
Brief Title: Evaluating Stress Response and Anxiety Score in Paediatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Huda Zainal Abidin, Lecturer and Anaesthetist, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A82010307
Record Dates: First submitted 2020-08-04; First posted 2020-08-26 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Anxiety and Fear; Anesthesia
Keywords: Paediatric; Intranasal; General anaesthesia; Dexmedetomidine; Anxiety score; cortisol
MeSH Terms: conditions — Anxiety Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Randomization of paediatric patients for general anaesthesia one arm: Intranasal dexmedetomidine another arm: Intranasal normal saline (placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Intranasal dexmedetomidine 1mcg/kg
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Intranasal normal saline equivalent to (1mcg/kg dose of dexmedetomidine)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Evaluating anxiety score in both arms
  Arms: Dexmedetomidine
Drug: Placebo — Evaluating anxiety score in both arms
  Arms: Placebo

SUMMARY:
To date, there have been no studies done relating serum cortisol levels and intranasal dexmedetomidine sedation. However, there was a behavioral study done on pediatric patients confirming reduction serum cortisol levels with perioperative dialogue intervention.There have been a number of studies done on adult patients indicating that dexmedetomidine was indeed capable of reducing level of anxiety with evidence of lower serum cortisol levels. Hence, we postulated that intranasal dexmedetomidine administration in pediatric patients will lower the serum cortisol levels but we need to evaluate the extent of reduction.

DETAILED DESCRIPTION:
Justification of study

With increase in number of pediatric patients undergoing surgery, efforts need to be placed on improving quality of perioperative care and patient comfort Intranasal administration of sedative agents will be far more comfortable and create a better environment for patients as most children have a fear of needles and may resist intravenous drug administration Intranasal administration is also a far simpler and less time-consuming technique with good bioavailability of administered drugs Reduction in postoperative analgesia requirement will result in early return to daily life activities, early discharge and overall reduced length of stay and hospital costs

Pre and intraoperative

All perioperative data will be collected by an investigator who is blinded to the patient's allocation. Once the caregiver has agreed and consented to participate in this study, upon admission (1 day prior to scheduled surgery) a baseline serum cortisol level will be taken concurrent with IV line setting and blood investigations. The fasting time for all patients will be at least 6 hours prior to surgery with clear fluids being allowed up to 2 hours prior to surgery.

On the day of surgery, the patient and caregiver will be called upon 1 hour prior to operating time and baseline hemodynamic parameters will be recorded (blood pressure, heart rate and pulse oximetry SpO2). Baseline Modified Yale Preoperative Anxiety Scale (m-YPAS) will be used as an assessment tool for measuring level of preoperative anxiety.

Baseline Modified Yale Preoperative Anxiety scale (m-YPAS) is an established and recognized tool for assessment of pediatric anxiety levels preoperatively. It is an observational checklist each consisting of four to six distinct behavioral descriptions. Four categories of behavior are assessed: activity, vocalizations, emotional expressivity, and state of apparent arousal. Partial weights are used to calculate a total score ranging from 23 (low anxiety) to 100 (high anxiety). Previous research has shown good to excellent inter and intra-observer reliability and validity.

Once the baseline parameters have been recorded, patient will receive the medication previously assigned via randomization delivered via mucosal atomizer device (MAD). Drugs will be administered by anesthetist or anesthetic medical officer only in safe setting with drugs for resuscitation and monitoring equipment available. They will be briefed on the workflow and timing of drug administration accordingly. The person responsible for delivering the medication will be blinded.

Hemodynamic parameters will be charted at 10 minutes intervals after the study medications have been served. Rescue drugs IV atropine 10 - 20mcg/kg will be given if the patient develops bradycardia (less than 2SDs for age) and fluid boluses if blood pressure drops to more than 20% of baseline or below 2SD of blood pressure for age.

2nd Modified Yale Preoperative Anxiety Scale (m-YPAS) will be assessed 10 minutes after delivering the study medications. This is followed by sedation score after 30 minutes and 3rd. m-YPAS if indicated.

Sedation and behavior score is a simplified scoring system that is based on observational charting. It comprises of 2 domains ranging from alert, awake, crying and resisting to asleep and not responding to mild prodding or shaking while being calm and cooperative. Higher scores indicate a higher level of sedation and are more favorable.

Once the patient has arrived in the operation theatre, the SpO2 monitoring probe will be attached and intravenous induction is carried out with IV Propofol 4 - 5mg/kg. This is followed by applying other standard monitoring appliances such as blood pressure cuff and ECG electrodes. IV fentanyl 1-2mcg/kg to obtund the laryngeal reflex and paralysis with IV esmeron 0.6-1mg/kg. Appropriate size endotracheal tubes (ETT) or laryngeal mask airway (LMA) will be inserted accordingly to secure the airway.

2nd sample of serum cortisol level will be taken within 10 minutes of induction of anesthesia. Maintenance of anesthesia with sevoflurane aiming at 1.0 minimum alveolar concentration (MAC). Intravenous fluid will be replaced according to (Holiday Segar Formula) using either HM solution or sterofundin.

IV paracetamol 15mg/kg will be given pre-emptively, followed by IV morphine 0.1mg/kg. IV Fentanyl boluses 0.5-1mcg/kg will be served if required based on the hemodynamic parameters.

Postoperative

Postoperatively patient will be monitored in recovery room for 30 minutes and pain will be assessed using Wong Baker Faces pain rating scale/FLACC for smaller children. Rescue analgesic IV Fentanyl 0.5-1mcg/kg will be given if required. The total requirement of IV Fentanyl and the discharge time will be recorded for reference.

Wong Baker Faces scale is tool created with children to help them communicate their pain. Now the scale is used around the world with people ages 3 and older, facilitating communication and improving assessment so pain management can be addressed accordingly. There are 6 faces with each face representing a person who has no pain (hurt), or some, or a lot of pain. The patient chooses the face that best depicts the pain they are experiencing.

The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. It is an observational based scale. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2. Higher scores indicate higher pain.

Statistical Analysis

The analyses will be performed using the IBM SPSS Statistics for Windows Version 21.0. The data will be manually entered into the software before the cleaning process takes place. The cleaning process is crucial to prevent any errors that may skew the results. After that, the actual analysis process will be carried out. In this study, descriptive statistics will be employed for selected variables. The findings will be presented based on the types of data and their distribution. Categorical Data, will be presented as frequencies and percentage. Numerical Data will be presented as means and standard deviations if normally distributed, and if not, as medians and interquartile ranges.

Comparison of Numerical Data between two independent groups that are normally distributed will be analyzed using the Independent t-test, while Mann-Whitney test will be used if the data for two independent groups are not normally distributed.

Hemodynamic parameters measurement (objective 3) will be analyzed using repeated measures ANOVA while Friedman test will be used if the Numerical Data are not normally distributed. All probability values are two-sided, and a level of significance of less than 0.05 (p-value < 0.05) will be considered as statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients age 1-12 years old
* Weight of patient between 10 - 60 kgs
* American Society of Anesthesiologist (ASA) I or II
* Scheduled for elective and emergency surgeries
* Caregivers able to understand and provide informed consent

Exclusion Criteria:

* Allergy to study drugs (dexmedetomidine, morphine, paracetamol etc.)
* Special need Children (Cerebral palsy, down syndrome, ADHD, ASD)
* Serious cardiac/respiratory diseases.
* Children with neuromuscular disorders or neurological diseases (epilepsy etc)
* Children with Metabolic disorders
* Difficult airway cases
* Children on any kind of steroid therapy / HPA diseases

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluating stress response | Baseline: (before giving study drugs) and 1 to half an hour after drugs given
  Evaluating stress response by measuring serum cortisol level (nmol/L)
Evaluating anxiety score | Baseline:(before giving study drugs) and 1 to half an hour after drugs given
  To compare mean anxiety score using modified Yale Preoperative Anxiety Scales (m-YPAS)

SECONDARY OUTCOMES:
Safety profile of Intranasal Dexmedetomidine in paediatric patients | Baseline and 10 minutes interval after study drugs given
  Monitoring the haemodynamic parameters (blood pressure in mmHg)
Safety profile of Intranasal Dexmedetomidine in paediatric patients | Baseline and 10 minutes interval after study drugs given
  Monitoring the haemodynamic parameters (heart rate in beats per minute)
Safety profile of Intranasal Dexmedetomidine in paediatric patients | Baseline and 10 minutes interval after study drugs given
  Monitoring the haemodynamic parameters (Oxygen saturation in percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Huda Zainal Abidin, MD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No
IPD will be considered for sharing if the the data is to be used for related study

REFERENCES:
- [Background] Isik B, Arslan M, Tunga AD, Kurtipek O. Dexmedetomidine decreases emergence agitation in pediatric patients after sevoflurane anesthesia without surgery. Paediatr Anaesth. 2006 Jul;16(7):748-53. doi: 10.1111/j.1460-9592.2006.01845.x. PMID 16879517
- [Background] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Background] Yuen VM, Hui TW, Irwin MG, Yao TJ, Chan L, Wong GL, Shahnaz Hasan M, Shariffuddin II. A randomised comparison of two intranasal dexmedetomidine doses for premedication in children. Anaesthesia. 2012 Nov;67(11):1210-6. doi: 10.1111/j.1365-2044.2012.07309.x. Epub 2012 Sep 5. PMID 22950484
- [Background] Yuen VM, Hui TW, Irwin MG, Yao TJ, Wong GL, Yuen MK. Optimal timing for the administration of intranasal dexmedetomidine for premedication in children. Anaesthesia. 2010 Sep;65(9):922-9. doi: 10.1111/j.1365-2044.2010.06453.x. PMID 20645951
- [Background] Akin A, Bayram A, Esmaoglu A, Tosun Z, Aksu R, Altuntas R, Boyaci A. Dexmedetomidine vs midazolam for premedication of pediatric patients undergoing anesthesia. Paediatr Anaesth. 2012 Sep;22(9):871-6. doi: 10.1111/j.1460-9592.2012.03802.x. Epub 2012 Jan 23. PMID 22268591